CLINICAL TRIAL: NCT00765167
Title: Training and Calibration of Dental Examiners
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: William DeVizio/VP - Clinical Research, Colgate Palmolive
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ATO-2007-PLA-01-RR
Record Dates: First submitted 2008-09-23; First posted 2008-10-02 (Estimated); Last update posted 2008-10-03 (Estimated); Status verified 2008-10

CONDITIONS: Dental Plaque
MeSH Terms: conditions — Dental Plaque | interventions — Fluorides; Triclosan; chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Placebo Comparator)
  Interventions: Drug: Fluoride
- B (Active Comparator)
  Interventions: Drug: Triclosan; Drug: Fluoride
- C (Active Comparator)
  Interventions: Drug: Chlorhexidine gluconate

INTERVENTIONS:
Drug: Fluoride — Brush half mouth twice daily for four days
  Arms: A
Drug: Triclosan — Brush half mouth daily for four days
  Arms: B
Drug: Chlorhexidine gluconate — Mouth rinsing with 15 ml for 30 seconds twice a day for four days
  Arms: C
Drug: Fluoride — Brush half mouth daily for four days
  Arms: B

SUMMARY:
Training and calibration of dental examiners

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers 18-65 years of age
* Good general health
* Must sign informed consent form
* Minimum of 20 natural uncrowned teeth (excluding third molars) must be present.
* No history of allergy to personal care consumer products, or their ingredients, relevant to any ingredient in the test products as determined by the dental/medical professional monitoring the study.

Exclusion Criteria:

1. Subjects unable or unwilling to sign the informed consent form.
2. Medical condition which requires pre-medication prior to dental visits/procedures
3. Moderate or advanced periodontal disease or heavy dental tartar (calculus).
4. 2 or more decayed untreated dental sites at screening.
5. Other disease of the hard or soft oral tissues.
6. Impaired salivary function (e.g. Sjogren's syndrome or head and neck irradiation).
7. Use of medications that can affect salivary flow (e.g. anticholinergics, adrenergics, antihistamines, vasoconstrictors or decongestants).
8. Use of antibiotics or antimicrobial drugs within 30 days prior to study visit #1.
9. Pregnant or nursing women.
10. Participation in any other clinical study within 1 week prior to enrollment into this study.
11. Allergy to chlorhexidine
12. Use of tobacco products
13. Subjects who must receive dental treatment during the study dates.
14. Current use of Antibiotics for any purpose.
15. Presence of an orthodontic appliance.
16. History of allergy to common dentifrice ingredients.
17. Immune compromised individuals (HIV, AIDS, immuno suppressive drug therapy)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-11; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Dental plaque | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Deasy, DDS, Principal Investigator
Locations (1):
- UMDNJ Dental School, Newark, New Jersey, United States